CLINICAL TRIAL: NCT01592162
Title: Dose-effect of Propofol for Anesthetic Induction: Double-blind Comparison of Different Propofol Formulations Administered Alone or With Remifentanil
Brief Title: Comparison of Different Propofol Formulations With or Without Remifentanil
Acronym: PropofolRemi
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011/34; 2011-002644-27 (Other: ANSM)
Record Dates: First submitted 2012-04-17; First posted 2012-05-07 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Anesthesia
MeSH Terms: interventions — Propofol; Sodium Chloride; Remifentanil; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- propofol 1% (Astra-Zeneca) - remi 0 (Active Comparator): propofol 1% (Astra-Zeneca)plus remifentanil 0 ng/ml
  Interventions: Drug: Propofol (Astra-Zeneca), NaCl 0.9%
- propofol 1% (Astra-Zeneca) - remi 2 (Active Comparator): propofol 1% (Astra-Zeneca)plus remifentanil 2 ng/ml
  Interventions: Drug: propofol 1% (Astra-Zeneca) and remifentanil
- propofol 1% (Astra-Zeneca) - remi 4 (Active Comparator): propofol 1% (Astra-Zeneca)plus remifentanil 4 ng/ml
  Interventions: Drug: propofol 1% (Astra-Zeneca) and remifentanil
- propofol 1% (Fresenius) - remi 0 (Active Comparator): propofol 1% (Fresenius) plus remifentanil 0 ng/ml
  Interventions: Drug: Propofol (Astra-Zeneca), NaCl 0.9%
- propofol 1% (Fresenius) - remi 2 (Active Comparator): propofol 1% (Fresenius) plus remifentanil 2 ng/ml
  Interventions: Drug: Propofol (Astra-Zeneca) and remifentanil
- propofol 1% (Fresenius) - remi 4 (Active Comparator): propofol 1% (Fresenius) plus remifentanil 4 ng/ml
  Interventions: Drug: Propofol (Astra-Zeneca) and remifentanil
- propofol 1% (B-Braun) - remi 0 (Active Comparator): propofol 1% (B-Braun) plus remifentanil 0 ng/ml
  Interventions: Drug: Propofol (B-Braun) and NaCl 0.9%
- propofol 1% (B-Braun) - remi 2 (Active Comparator): propofol 1% (B-Braun) plus remifentanil 2 ng/ml
  Interventions: Drug: Propofol (B-Braun) and remifentanil
- propofol 1% (B-Braun) - remi 4 (Active Comparator): propofol 1% (B-Braun) plus remifentanil 4 ng/ml
  Interventions: Drug: Propofol (B-Braun) and remifentanil

INTERVENTIONS:
Drug: Propofol (Astra-Zeneca), NaCl 0.9% — propofol administered by a closed-loop system and saline
  Arms: propofol 1% (Astra-Zeneca) - remi 0
Drug: propofol 1% (Astra-Zeneca) and remifentanil — propofol administered by a closed-loop system and remifentanil (2 ng/ml, target controled infusion)
  Arms: propofol 1% (Astra-Zeneca) - remi 2
Drug: propofol 1% (Astra-Zeneca) and remifentanil — propofol administered by a closed-loop system and remifentanil (4 ng/ml, target controled infusion)
  Arms: propofol 1% (Astra-Zeneca) - remi 4
Drug: Propofol (Astra-Zeneca), NaCl 0.9% — propofol administered by a closed-loop system and saline
  Arms: propofol 1% (Fresenius) - remi 0
Drug: Propofol (Astra-Zeneca) and remifentanil — propofol administered by a closed-loop system and remifentanil (2 ng/ml, target controled infusion)
  Arms: propofol 1% (Fresenius) - remi 2
Drug: Propofol (Astra-Zeneca) and remifentanil — propofol administered by a closed-loop system and remifentanil (4 ng/ml, target controled infusion)
  Arms: propofol 1% (Fresenius) - remi 4
Drug: Propofol (B-Braun) and NaCl 0.9% — propofol administered by a closed-loop system and saline
  Arms: propofol 1% (B-Braun) - remi 0
Drug: Propofol (B-Braun) and remifentanil — propofol administered by a closed-loop system and remifentanil (2 ng/ml, target controled infusion)
  Arms: propofol 1% (B-Braun) - remi 2
Drug: Propofol (B-Braun) and remifentanil — propofol administered by a closed-loop system and remifentanil (4 ng/ml, target controled infusion)
  Arms: propofol 1% (B-Braun) - remi 4

SUMMARY:
The objective of this study is to evaluate the influence of different propofol formulations (plain or with remifentanil) on anesthetic induction. Propofol plain or with remifentanil is administered using a closed-loop algorithm in order to reach a Bispectral Index target of 50.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for an intravenous induction of anesthesia with propofol

Exclusion Criteria:

* Age under 18
* Pregnancy or breastfeeding
* Allergy to propofol, soya or peanuts,
* Allergy to remifentanil,
* History of central neurological disorder or brain injury,
* Patients receiving psychotropic drugs,
* Patient with a pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2013-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
necessary dose of propofol to obtain the induction of anesthesia (defined by a bispectral index < 60 over 30 continuous seconds) | one hour after anesthesia

SECONDARY OUTCOMES:
calculated concentrations of propofol at the end of the anesthetic induction | one hour after anesthesia
pain at injection | one hour after anesthesia
heart rate modifications induced by anesthetic induction | one hour after anesthesia
patient's satisfaction | one day after anesthesia
arterial pressure modifications induced by anesthetic induction | one hour after anesthesia
Disappearance of the eyelash reflex | One hour after anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Study Chair — Hopital Foch
Locations (2):
- France (2):
  - CHU Besançon, Besançon
  - Hopital Foch, Suresnes, Île-de-France Region